CLINICAL TRIAL: NCT06994429
Title: Exploring the Application Value of New Magnetic Resonance Imaging Technologies in Non-invasive Quantitative Assessment of Graft Function After Liver Transplantation
Status: Enrolling by invitation | Type: Observational
Sponsor: Zhen Li (Other)
Responsible Party: Sponsor-Investigator, Zhen Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202411026
Record Dates: First submitted 2025-04-23; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Liver Transplantation; MRI; Graft Function
Keywords: Graft Function; Liver Transplantation; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: MRI Techniques for Graft Function Assessment — ### Intervention Description
  The intervention in this study is the use of advanced MRI techniques for assessing liver transplant graft function. It includes:
  * **Diffusion Weighted Imaging (DWI):** To evaluate tissue integrity and detect early graft dysfunction.
  * **Dynamic Contrast-Enhanced MRI (DCE-MRI):** To assess vascular complications and blood flow in the graft.
  * **Blood Oxygenation Level-Dependent (BOLD) MRI:** To monitor oxygenation levels, indicative of graft health.
  These MRI methods provide a non-invasive, comprehensive assessment of liver graft function, distinguishing this intervention from traditional invasive methods like biopsy.

SUMMARY:
Title: Exploring the Application Value of New Magnetic Resonance Imaging Technologies in Non-invasive Quantitative Assessment of Graft Function after Liver Transplantation

Purpose of the Study:

This study aims to investigate the value of new imaging technologies in assessing early graft function in patients who have undergone liver transplantation. By analyzing clinical, imaging, laboratory, and pathological data from liver transplant patients, the study seeks to establish a non-invasive method for diagnosing, evaluating treatment efficacy, and predicting outcomes related to graft function.

Background:

Liver transplantation is a critical treatment for end-stage liver disease and acute liver failure. While it significantly improves patients' quality of life and survival rates, complications such as graft dysfunction can occur post-surgery. Traditional methods for assessing graft function, including liver function tests, imaging studies (like ultrasound and CT), and biopsy, have limitations in sensitivity and specificity. Therefore, there is a need for safer, non-invasive techniques that can provide a comprehensive assessment of graft function.

Study Design:

Type: Prospective study Participants: 1000 liver transplant patients who meet specific inclusion criteria, such as undergoing MR imaging post-transplant.

Exclusion Criteria: Patients with contraindications for MRI, such as implanted devices or claustrophobia.

Methods:

Participants will undergo MRI scans using advanced techniques like diffusion-weighted imaging (DWI) and dynamic contrast-enhanced MRI (DCE-MRI) to evaluate graft function. Clinical and laboratory data will also be collected for comprehensive analysis.

Potential Benefits:

This study aims to enhance the early detection of graft dysfunction, allowing for timely interventions that could improve patient outcomes and prolong graft survival.

Risks and Safeguards:

While there is a risk of privacy breaches regarding patient data, all information will be handled confidentially and used solely for research purposes. Patient identities will be protected throughout the study.

Conclusion:

The findings from this study could lead to improved non-invasive assessment methods for liver transplant patients, ultimately enhancing clinical decision-making and patient care.

DETAILED DESCRIPTION:
Title: Exploration of New Magnetic Resonance Imaging Technologies for Non-invasive Quantitative Assessment of Graft Function after Liver Transplantation

Principal Investigator: Professor Li Zhen

Research Institution: Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology

Objective:

The study aims to explore the value of new imaging technologies in assessing the early postoperative graft function in liver transplant patients. It seeks to establish relationships between imaging parameters, body composition, metabolic diseases, and graft function, with the goal of guiding clinical treatment and improving survival rates and quality of life for liver transplant patients.

Study Design:

Type: Prospective Sample Size: 1000 cases, calculated based on multivariate analysis requirements and considering a dropout rate of around 20%.

Eligibility Criteria:

Inclusion: Patients who have undergone liver transplantation and are scheduled for MR examinations.

Exclusion: Patients with contraindications for MRI such as pacemakers, unknown metallic implants, neurostimulators, claustrophobia, or those who cannot hold their breath for the duration of the MR scan.

Withdrawal Criteria:

Serious adverse events Poor compliance Patient's request to withdraw Investigator's decision that continuation of the study is not in the patient's best interest

Study Process:

Imaging Data Collection: Patients meeting the criteria will be informed and consented. They will undergo MR scans after fasting for 8 hours and hydrating for 4 hours. Imaging data will be collected and documented.

Imaging Data Processing: DICOM format images will be copied from the PACS system and analyzed using imaging processing software to record relevant parameters.

Clinical Data Collection: Clinical and laboratory data will be collected through the RIS system at Tongji Hospital, including liver function tests, blood tests, and pathological data. Patient histories and treatment information will also be documented.

Risks and Precautions:

Risks: Potential of patient privacy due to the use of imaging and electronic medical records.

Precautions: All data used in the study will be anonymized to protect patient identity and will not be used for commercial purposes.

Data Collection and Statistical Analysis:

Data will be analyzed using statistical software like SPSS after collection and organization of clinical, laboratory, and outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone liver transplantation.
2. Patients who are scheduled for MR imaging post-transplant.
3. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. Patients with contraindications for MRI, such as pacemakers, unknown metallic implants, or neurostimulators.
2. Patients with claustrophobia or inability to tolerate the required breath-holds for MRI.
3. Patients who cannot comply with the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes post-liver transplant patients at Tongji Hospital who are eligible for MRI scans and meet the inclusion and exclusion criteria. Participants are of all ages and genders, ensuring a broad demographic representation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Exploring the Application Value of New Magnetic Resonance Imaging Technologies in Non-invasive Quantitative Assessment of Graft Function after Liver Transplantation | The study is a prospective analysis of 1000 liver transplant patients to assess graft function using MRI. The study is expected to last up to 5 years.
  This study focuses on employing advanced MRI techniques to non-invasively evaluate the function of liver transplant grafts, distinguishing it from traditional methods by offering a comprehensive, less invasive approach to post-transplant care.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, NO.1095 jiefang avenue, Wuhan, Hubei, China